CLINICAL TRIAL: NCT03164187
Title: Evaluation of Type 2 Diabetes Treatment in AZERbaijan
Brief Title: Evaluation of Type 2 Diabetes Treatment
Status: Completed | Type: Observational
Sponsor: Servier Affaires Médicales (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Other Study IDs: EDIAZER
Record Dates: First submitted 2017-04-12; First posted 2017-05-23 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabeton MR 60
  Interventions: Drug: Diabeton 60 MR

INTERVENTIONS:
Drug: Diabeton 60 MR — Administer Diabeton MR 60 mg 1/2 tablet. Increasing dosage of Diabeton MR 60 mg by ½ tablet is recommended if fasting glucose level exceeds 6 mmol/L.

SUMMARY:
The aim of this study is to analyze the efficacy of Diabeton 60 MR as intensive sugar-lowering therapy into routine clinical practice, in patients for whom the treating physician has already decided to prescribe this medication. This concerns untreated newly diagnosed patients uncontrolled by diet, and patients uncontrolled by metformin.

ELIGIBILITY:
Inclusion Criteria:

- Type 2 diabetes patients:

* Males and females, aged over 35
* Currently treated: with diet only, or with metformin therapy for at least 3 months prior to inclusion
* Who have not been able to achieve target level of glycaemia, with glycated hemoglobin (HbA1c) level exceeding 7%.

Exclusion Criteria:

Patients with at least one of the following criteria are not included in the study:

* Type 1 diabetes
* Severe liver (ALT and AST levels 2.5 times as high as upper level of normal range) or renal insufficiency (creatinin plasma level above 140 µmole/L)
* Patients who are on insulin therapy, or at risk to receive an insulin treatment in the next 4 months, according to physician judgment.
* Intolerance to Gliclazide if such prescription was done in the past
* Pregnancy and breast-feeding
* Night workers or patients able to skip meals
* Presence of any contraindication listed in the SmPC.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-06-10 (Actual)

PRIMARY OUTCOMES:
Decrease in HbA1c | over 4 months
Percentage of patients achieving HbA1c level ≤ 7 % | week 16.

SECONDARY OUTCOMES:
number of hypoglycemia episodes | Week 0, 2, 4, 6, 8 and week 16.
Mean daily dosage of Diabeton MR | Week 2, 4, 6, 8 and 16

CONTACTS AND LOCATIONS:
Locations (4):
- Azerbaijan (4):
  - Azerbaijan Republic Ministry of Health Republic Endocrinology Center, Baku
  - Azer-Turk Med clinic, Baku
  - Hospital of oil workers, polyclinics and private clinics, Baku
  - Medical Clinic of Azerbaijan Medical University, Baku

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- [Background] Mirzazada VA, Huseynova RA, Mustafayeva SA, Gasimova FN, Ahmadova U, Ismayilova N, Kerimova V, Mehdiyeva H, Suleymanova R, Maharramova Z, Iskandarli G, Gurbanova O, Aghayeva S, Malikova S, Ismayilova K, Salimkhanova K. Evaluation of Type 2 Diabetes Treatment with Gliclazide Modified Release in Azerbaijan (the EdiAzer study): Results from a 16-Week Observational Clinical Study. J Diabetol. 2020 Sep-Dec;11(3):175-182. doi: 10.4103/JOD.JOD_5_20
- See also: Scientific publication — http://www.journalofdiabetology.org/article.asp?issn=2078-7685;year=2020;volume=11;issue=3;spage=175;epage=182;aulast=Mirzazada;type=0